CLINICAL TRIAL: NCT03726697
Title: Effect of Tahneek With Dates on Hypoglycemia in Newborn Infants: A Randomised Control Trial
Brief Title: Effect of Tahneek on Hypoglycemia in Newborn Infants
Acronym: THIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Principal Investigator, Jubara Alallah, Assistant Professor of Pediatrics, King Abdullah International Medical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KAIMRC
Record Dates: First submitted 2018-10-30; First posted 2018-10-31 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Neonatal Hypoglycemia; Infant, Small for Gestational Age; Macrosomia, Fetal; Intrauterine Growth Restriction; Premature Infant; Neonatal; Hypoglycemia, Diabetes, Maternal
Keywords: Tahneek; Neonatal; Hypoglycemia, Diabetes, Maternal; Neonatal Hypoglycemia; late preterm infants; Prevention; IUGR
MeSH Terms: conditions — Fetal Macrosomia; Fetal Growth Retardation; Premature Birth; Hypoglycemia; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Parents and Statistician are blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tahneek (Experimental): Infants receiving a single dose of soft date, prepacked by the pharmacy containing glucose equivalent to 200mg/kg at 1 hour after birth in the nursery.
  Interventions: Other: Tahneek
- CONTROL (No Intervention): Infants at risk for transient neonatal hypoglycemia following standard-of-care.

INTERVENTIONS:
Other: Tahneek — A single dose of soft date containing glucose equivalent to 200mg/kg at 1 h after birth will be massaged into the buccal mucosa of the palate and cheek from right to left side, until the date paste is fully absorbed
  Arms: Tahneek

SUMMARY:
Tahneek is an Arabic word which means putting something sweet such as dates, in the infant's mouth after the birth. Neonatal hypoglycemia is common in the first few days after birth. Up to 15 % of normal newborn babies will have low blood glucose concentrations. It has been demonstrated that treatment of neonatal hypoglycemia with oral dextrose gel was more effective than feeding alone in reversing the hypoglycemia, and also reduced the rate of NICU admission. investigators study is using dates to asses its effect on hypoglycemia in infants at risk.

DETAILED DESCRIPTION:
Tahneek is an Arabic word which means putting something sweet such as dates, in the infant's mouth after the birth. It is a noble practice in Islam, with which the newborn is greeted upon entering into life, usually before milk feeds. It is done by rubbing a softened date on the palate of the new-born just after the birth. The tahneek also exercises the muscles of the mouth and helps with the circulation of blood in the mouth - this may help the baby to be able to suck and take mother's milk. Neonatal hypoglycemia is common in the first few days after birth. Up to 15 % but the incidence in babies with risk factors is much greater upto 50 % in infants of diabetic mothers, large and small babies and 66 % in preterm babies. Neonatal hypoglycemia is associated with brain damage, death and developmental delay in later life. Treatment of neonatal hypoglycemia with oral dextrose gel was more effective than feeding alone in reversing hypoglycemia, and thus reducing the rate of NICU admission for hypoglycemia. investigators study is using dates to asses its effect on hypoglycemia in infant at risk.

ELIGIBILITY:
Inclusion Criteria:

* Babies at risk of hypoglycemia less than 1 hour old admitted to the normal nursery.
* Infants of diabetic mothers (any type of diabetes)
* Late Preterms (34 - 37 weeks' gestation)
* Low birth weight (< 2.5 kg ) or Small for gestational age
* Large for gestational age (> 4 kg or > 90th centile on Fenton's growth chart)

Exclusion Criteria:

* Major congenital abnormality including severe cleft lip and palate.
* Babies requiring NICU admission immediately after birth
* Babies less than 34 weeks of age.
* Babies whose parents refused to consent

Max Age: 1 Hour | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 324 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
Hypoglycemia | first 48 hours of life
  infants who meet eligibility criteria and parents have consented will receive a single dose of soft date, prepacked by the pharmacy containing glucose equivalent to 200mg/kg within 1 h after birth. Assess glucose level after 1 feed compared to controls with similar risk factors who are not received Tahneek. hypoglycemia defined as any blood glucose concentration < 2.6 mmol/L.
Admission to NICU for hypoglycemia | first 48 hours of life
  infants at-risk will be followed to measure NICU admission data and glucose values during hospitalization.

SECONDARY OUTCOMES:
Hyperglycemia | 48 hours
  infants at-risk who received Tahneek will be followed until hospital discharge to measure NICU admission data and glucose values during hospitalization. hyperglycemia defined as any blood glucose concentration > 10 mmol/L.
Breastfeeding | 6 months
  will asses the breastfeeding rate in the study infants, compared to controls at discharge from hospital (full or exclusive) and at 6months of age.
Pain scale | 48 hours
  Pain scale as measured by Neonatal intensive pain scale during the first 48 hrs of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Jubara Alallah, MD, Principal Investigator — King Abdullah International Medical Research Center
Locations (1):
- King Abdulaziz Medical City, Jeddah, WR, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided